CLINICAL TRIAL: NCT05166798
Title: Establishing a Dose-response Relationship for the Effects of a Cognitive Control Training on Depression Vulnerability
Brief Title: Optimal Dose of a Cognitive Control Training for Depression Vulnerability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BC-10551
Record Dates: First submitted 2021-11-10; First posted 2021-12-22 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Major Depression in Remission
Keywords: Depression; Remission; Relapse prevention; Cognitive control training; Internet intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Cognitive control training: The adaptive Paced Auditory Serial Addition Task (aPASAT) is a Cognitive Control Training where participants need to click on the sum of the last two heard digits. Task difficulty is modified based on the participants' current task performance, allowing training of cognitive control. Five intervention groups will each receive a different amount of sessions.
  Interventions: Behavioral: Cognitive control training
- Control group (No Intervention): Waitlist control group: Participants randomized to the control group will not perform the cognitive control training during the study, but will be given the opportunity to follow the training afterwards.

INTERVENTIONS:
Behavioral: Cognitive control training — The five intervention groups will receive either 1, 5, 10, 15 or 20 training sessions with the Adaptive Paced Auditory Serial Addition Task (aPASAT).
  Arms: Intervention group

SUMMARY:
This study aims to examine the dose-response relationship of an online adaptive cognitive control training on depressive symptomatology and rumination. Participants will be randomized over six groups, each receiving a different dose (0, 1, 5, 10, 15 or 20 sessions) of a cognitive control training in remitted depressed patients. An adaptive Paced Auditory Serial Addition Task will be used as cognitive control training.

DETAILED DESCRIPTION:
Depression is often associated with cognitive impairments and recent studies have found that for some people, these cognitive problems persist after remission of depression. These cognitive impairments could be a risk factor for recurrence of depressive episodes. Cognitive control training aims to address these cognitive impairments and decrease the risk of recurrence of depression.

One promising operationalization of cognitive control training is the adaptive Paced Auditory Serial Addition Task, but currently, it's unclear how many sessions one should complete in order to obtain cognitive- and emotional transfer effects. By comparing multiple groups with a different number of sessions (0, 1, 5, 10, 15 and 20), with measures at post (one month after baseline) and two follow-up periods (at 3 months and 6 months after baseline), this study examines the effects of an online cognitive control training on depressive vulnerability factors.

ELIGIBILITY:
Inclusion Criteria:

* History of ≥ 1 depressive episode(s)
* Currently in remission (≥ 3 months)
* Access to a computer with an internet connection

Exclusion Criteria:

* Ongoing depressive episode
* Psychotic disorder (current and/or previous)
* Neurological impairments (current and/or previous)
* Excessive substance abuse (current and/or previous)
* Use of antidepressant medication is allowed if kept at a constant level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory (BDI-II-NL) | baseline, post training (one month after baseline), 3 month follow-up after baseline, 6 month follow-up after baseline
  Self-report questionnaire with 21 items, depression symptom severity, scores can range from 0 to 63, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Change in Perseverative Thinking Questionnaire (PTQ-NL) | baseline, post training (one month after baseline), 3 month follow-up after baseline, 6 month follow-up after baseline
  Change from baseline in perseverative thinking. The PTQ-NL consist of 15 items and are assessed using scores ranging from 0 (never) to 4 (almost always). Lower scores indicate lower levels of preservative thinking.
Change in Cognitive Emotion Regulation Questionnaire (CERQ) | baseline, post training (one month after baseline), 3 month follow-up after baseline, 6 month follow-up after baseline
  Self-reported measure for emotion regulation: a 36-item questionnaire, consisting of 9 subscales (Self-blame, Other-blame, Rumination, Catastrophizing, Putting into Perspective, Positive Refocusing, Positive Reappraisal, Acceptance and Planning). Each item is rated on a 1 to 5 scale (1 = almost never and 5 = almost always). Higher subscale scores represent more frequent use of a specific cognitive strategy.
Change in Adult Temperament Questionnaire (ATQ), Effortful Control subscale | baseline, post training (one month after baseline), 3 month follow-up after baseline, 6 month follow-up after baseline
  Measured by the subscale Effortful Control (EC) from the Adult Temperament Questionnaire (ATQ).
Change in Burnout Assessment Tool (BAT) | baseline, post training (one month after baseline), 3 month follow-up after baseline, 6 month follow-up after baseline
  The Burnout Assessment Tool (BAT) is used to assess burn-out risk. The score ranges from 1 to 5, with higher scores indicating a higher risk of burn-out.
Change in Remission from Depression Questionnaire (RDQ-NL) | baseline, post training (one month after baseline), 3 month follow-up after baseline, 6 month follow-up after baseline
  The Remission from Depression Questionnaire has 41 items, which assess domains such as positive mental health, life satisfaction, and sense of well-being. The items are scored 0 (not at all or rarely true), 1 (sometimes true) or 2 (often or almost always true).
Change in non-adaptive PASAT performance | baseline, post training (one month after baseline), 3 month follow-up after baseline, 6 month follow-up after baseline
  A non-adaptive computerized version of the Paced Auditory Serial- Addition Task (PASAT) was used as a measure of participants' working memory abilities. Higher accuracy scores suggest greater cognitive control resources.
Change in n-back performance | baseline, post training (one month after baseline)
  The n-back task is a classic cognitive working memory task during which participants are asked to decide if a digit appearing on a screen is the same as the digit that appeared n stimuli earlier (n-back).

OTHER OUTCOMES:
Change in List of Threatening Experiences (LTE-Q) | 3 month follow-up after baseline, 6 month follow-up after baseline
  In the LTE questionnaire, unpleased life events are listed and participants are asked if these events occurred recently. The LTE-Q contains 13 items for which "yes" or "no" are the two possible answers.
Change in Credibility and Expectancy Questionnaire (CEQ) | baseline, post training (one month after baseline)
  The 6-item CEQ measures ratings of treatment credibility, acceptability/satisfaction, and expectations for success.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Koster, Professor, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent, Oost-Vlaanderen
  - Ghent University, Ghent, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized individual participant data can be stored on Open-Science Framework (OSF).
Supporting Information: Analytic Code

REFERENCES:
- [Derived] Vander Zwalmen Y, Demeester D, Hoorelbeke K, Verhaeghe N, Baeken C, Koster EHW. The more, the merrier? Establishing a dose-response relationship for the effects of cognitive control training on depressive symptomatology. J Consult Clin Psychol. 2025 Mar;93(3):161-175. doi: 10.1037/ccp0000945. PMID 40014506
- [Derived] Vander Zwalmen Y, Hoorelbeke K, Demeester D, Koster EHW. High-Frequency Cognitive Control Training for Depression: Case Report. JMIR Form Res. 2024 Nov 29;8:e56598. doi: 10.2196/56598. PMID 39612206